CLINICAL TRIAL: NCT06969326
Title: Topical Estrogen: Brief Intervention to Improve Postoperative Experience for Transgender Men Undergoing Hysterectomy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Beth Cronin, Division Director, Division of General Obstetrics and Gynecology, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2255554-1
Record Dates: First submitted 2025-02-10; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Bleeding; Gender Dysphoria; Hysterectomy
Keywords: gender dysphoria; gender affirmation; hysterectomy
MeSH Terms: conditions — Postoperative Hemorrhage; Gender Dysphoria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Standard surgical treatment will be provided
  Interventions: Other: No intervention
- Estradiol (Experimental): Application of topical estradiol at conclusion of surgery
  Interventions: Drug: Use of topical estradiol

INTERVENTIONS:
Drug: Use of topical estradiol — The investigators will conduct a double blinded randomized control pilot trial. Participants will be randomized in 1:1 fashion to either receive no treatment or receive 2g of estradiol cream, placed after clearing the vaginal vault of any blood and discharge, at the conclusion of the surgery.
  Arms: Estradiol
Other: No intervention — This arm will not receive estradiol or other cream
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if applying a single dose of topical estrogen cream in the operating room at the end of your hysterectomy (removal of uterus and cervix) improves the postoperative experience with bleeding and potential symptoms of dysphoria (a feeling of discomfort or distress). Topical estrogen cream is sometimes used if patients have increased risk of bleeding with surgery but is not currently utilized in a consistent way. This study aims to answer the question of whether this is a helpful treatment and should be included in standard postoperative care.

DETAILED DESCRIPTION:
OBJECTIVES, SPECIFIC AIMS, BACKGROUND Vaginal bleeding causes significant dysphoria in many transgender men. The goal of hysterectomy for many patients is to eliminate the risk of bleeding, but the initial postoperative period often involves postoperative spotting and bleeding for patients, worsening the dysphoria around the time of surgery. Some patients have significant vaginal atrophy secondary to testosterone use, which is likely exacerbating this issue. Unfortunately, application of vaginal estrogen is messy and can worsen dysphoria symptoms for transgender individuals, making it not ideal for home use in the pre and postoperative periods.

Postoperative bleeding often prompts contacts with the health care system, especially when patients are experiencing dysphoria. These health system contacts are costly to patients, providers, and clinics particularly when the bleeding does not require intervention. Therefore, the investigators propose to pilot a trial of immediate postoperative intravaginal estrogen to prevent postoperative bleeding and decrease resulting health system contacts.

This pilot study will help to inform current practices about a novel process to decrease postoperative bleeding and dysphoria. This will help determine whether a simple intraoperative medication administration can improve the postoperative experience for patients and should help contribute data to guide future research in a patient population that has been under studied.

SIGNIFICANCE Bleeding related dysphoria is a common occurrence for many transmasculine individuals. A recent study of transgender adolescents demonstrated 93% had increased gender dysphoria or distress related to menses with many seeking care for menstrual management to achieve amenorrhea. (Schwartz 2022) Many patients achieve amenorrhea with initiation of testosterone and transgender patients are typically maintained on testosterone therapy for at least 6 months prior to gender affirming hysterectomy. Postoperative bleeding after hysterectomy, even in a well counseled patient, can be a dysphoric experience to manage in the postoperative period and impact patient satisfaction.

A recent study examined incidence and management of postoperative bleeding after gender affirming hysterectomy (GAH) which showed over 52% of the cohort called the clinic to report postoperative vaginal bleeding concerns. (Cipres 2023) Results showed that 88% had spotting or light bleeding requiring 1-2 pads per day in the first week after surgery. Patients who had had preoperative menstrual suppression had a higher (60%) frequency of postoperative bleeding concerns. Examinations revealed atrophy and granulation tissue as the source of bleeding. The authors hypothesize this was due to impaired tissue healing from the exogenous testosterone resulting in tissue friability and granulation tissue. (Cipres 2023) As vaginal bleeding could worsen gender dysphoria, these findings support the need for patient counseling on postoperative bleeding expectations and identification of interventions to reduce vaginal bleeding after GAH. Another recent retrospective study also demonstrated a higher rate of vaginal laceration during GAH compared to cisgender cohort (90% vs. 4.6%), along with increased use of electronic medical record (EMR) messages or calls for vaginal bleeding (27 vs 15%). (Pando 2024)

Cytopathology studies of hysterectomy and cervicovaginal specimens of patients on testosterone support the conclusion that testosterone exposure can induce histologic changes in the squamous epithelium of the cervix and vagina. (Khalifa 2019) While it is not proven if these changes impact wound healing, it may play a role in the healing process. Research investigating incidence of vaginal cuff dehiscence in GAH mostly demonstrates mixed results however one small study demonstrated that transgender individuals on testosterone may be at increased risk of cuff dehiscence. The authors hypothesize that changes in the vaginal epithelium may lead to poor wound healing which increases cuff dehiscence rates. (O'Connor 2023) Cuff dehiscence is a rare complication of laparoscopic hysterectomy which is why the focus of this study to examine patient reported quality of life measures after surgery.

Rahn et al. demonstrated that preoperative vaginal estrogen application for 6 weeks prior to vaginal surgery in women led to increased synthesis of mature collagen, decreased degradative enzyme activity and increased thickness of vaginal wall when looking at apical wall biopsies. This suggests that topical estrogen improves the substrate for suture placement at the time of surgery. (Rahn 2014) Additional studies demonstrated improved tissue quality markers postoperatively with administration of vaginal estrogen ring after pelvic reconstructive surgery. (Karp 2012) Finally, a recent study examined surgical outcomes after native tissue apical prolapse repair with perioperative estrogen versus placebo did not show reduced postoperative prolapse at 12 months but did show benefit of estrogen for reducing atrophy-related symptoms in the postoperative period. (Rahn 2023) Considering this, it is possible that postoperative vaginal estrogen could improve vaginal healing in patients using testosterone prior to their GAH and help reduce vaginal bleeding postoperatively.

Postoperative estrogen has limited data in gender diverse populations but presents as promising measure for decreasing postoperative dysphoria among transgender men.

Currently topical estrogen is given at the discretion of the surgeon in the postoperative period in transgender men. Patients are typically chosen if it appears that they have increased atrophy or small lacerations during surgery and estrogen cream is applied in the operating room. There are no evidence-based protocols to inform this decision or support the use of estrogen in this population. However, there is evidence demonstrating transgender patients have higher rates of clinic communication due to bleeding concerns. We aim to examine if a simple intraoperative application of estrogen will decrease postoperative bleeding and subsequent dysphoria. This study will contribute to the current literature and help to inform a future multicenter trial to address perioperative experiences for transgender individuals undergoing gender affirming hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Gender diverse/transgender men
2. Age 18 or older
3. Have been on testosterone for at least 6 months with plan to undergo gender-affirming hysterectomy and are willing to be randomized to the use of topical estrogen postoperatively.
4. Have stable physical and mental health
5. No contraindications to estrogen therapy
6. Must be proficient in English or Spanish
7. Must have access to a device to receive text messages for study follow up
8. Must agree to allow their medical data to be used for research purposes

Exclusion Criteria:

1. Under age 18
2. Have not been on testosterone for at least 6 months prior to planned hysterectomy
3. Known allergy to topical estrogen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of one-time topical estrogen application for reducing postoperative health system contacts for vaginal bleeding in the first two weeks post hysterectomy. | 2 weeks
  The investigators hypothesize that administration of postoperative estrogen cream vaginally in the operating room will decrease the need for health system contact for bleeding in the initial postoperative period.
  Patients will be asked to complete a brief email survey on postoperative days: 1, 3, 7, & 14 as well as at final postoperative visit ~42 days. This survey will target multiple things
  Outcome 1: Quantity of bleeding Determined by patient report: 1) small amount of spotting with wiping; 2) Staining pad, changing every 3-4 hours; 3) Bleeding like a light period; 4) Passing clots/heavy bleeding
  Additionally, chart review will be completed to assess for ED visits, office phone calls, MyChart Messages and any after-hours pages will be recorded.
Examine the impact of topical estrogen application on postoperative healing as defined by number of days of bleeding and patient Quality of Life Measures. | 6 weeks
  The investigators hypothesize that this intervention will demonstrate improved patient bleeding and dysphoria symptoms during the postoperative recovery period. The investigators will also measure mental health impact.
  Pre and postoperative Vanderbilt Mini Patient-Reported Outcome Measure - Gender (VMP-G)) scores will be obtained. This is a validated tool that assesses gender identity and gender affirming procedures as well as quality of life, self-concept, satisfaction, and gender dysphoria. (Hung 2023).

OTHER OUTCOMES:
Evaluate the efficacy of one-time topical estrogen application for reducing postoperative health system contacts for vaginal bleeding in the first two weeks post hysterectomy. | 2 weeks
  Additional outcomes:
  Outcome 2: Total days of postoperative bleeding (patient report) Outcome 3: Pain Scores on 0-10 scale at following intervals: postoperative days: 1, 3, 7, & 14 as well as at final postoperative visit ~42 days.
  Outcome 4: Types and doses of pain medication taken Outcome 5: Worsening dysphoria symptoms (yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- Women & Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schwartz BI, Effron A, Bear B, Short VL, Eisenberg J, Felleman S, Kazak AE. Experiences with Menses in Transgender and Gender Nonbinary Adolescents. J Pediatr Adolesc Gynecol. 2022 Aug;35(4):450-456. doi: 10.1016/j.jpag.2022.01.015. Epub 2022 Feb 3. PMID 35123055
- [Background] Rahn DD, Richter HE, Sung VW, Pruszynski JE, Hynan LS. Perioperative Vaginal Estrogen as Adjunct to Native Tissue Vaginal Apical Prolapse Repair: A Randomized Clinical Trial. JAMA. 2023 Aug 15;330(7):615-625. doi: 10.1001/jama.2023.12317. PMID 37581673
- [Background] Rahn DD, Good MM, Roshanravan SM, Shi H, Schaffer JI, Singh RJ, Word RA. Effects of preoperative local estrogen in postmenopausal women with prolapse: a randomized trial. J Clin Endocrinol Metab. 2014 Oct;99(10):3728-36. doi: 10.1210/jc.2014-1216. Epub 2014 Jun 20. PMID 24947034
- [Background] Pando C, Gerlach LR, Challa SA, Pan AY, Francis J. Operative Complications, Vaginal Bleeding, and Practice Considerations for Patients on Testosterone Undergoing Gender-Affirming Hysterectomy. J Minim Invasive Gynecol. 2024 Oct;31(10):836-842. doi: 10.1016/j.jmig.2024.05.026. Epub 2024 May 31. PMID 38823625
- [Background] Khalifa MA, Toyama A, Klein ME, Santiago V. Histologic Features of Hysterectomy Specimens From Female-Male Transgender Individuals. Int J Gynecol Pathol. 2019 Nov;38(6):520-527. doi: 10.1097/PGP.0000000000000548. PMID 30252728
- [Background] Karp DR, Jean-Michel M, Johnston Y, Suciu G, Aguilar VC, Davila GW. A randomized clinical trial of the impact of local estrogen on postoperative tissue quality after vaginal reconstructive surgery. Female Pelvic Med Reconstr Surg. 2012 Jul-Aug;18(4):211-5. doi: 10.1097/SPV.0b013e31825e6401. PMID 22777369
- [Background] Hung YC, Park BC, Assi PE, Perdikis G, Drolet BC, Kassis SA. Multidimensional Assessment of Patient-Reported Outcomes After Gender-Affirming Surgeries Using a Validated Instrument. Ann Plast Surg. 2023 Nov 1;91(5):604-608. doi: 10.1097/SAP.0000000000003652. Epub 2023 Aug 12. PMID 37553914
- [Background] Cipres DT, Shim JY, Grimstad FW. Postoperative Vaginal Bleeding Concerns after Gender-Affirming Hysterectomy in Transgender Adolescents and Young Adults on Testosterone. J Pediatr Adolesc Gynecol. 2023 Feb;36(1):33-38. doi: 10.1016/j.jpag.2022.09.002. Epub 2022 Sep 8. PMID 36089115